CLINICAL TRIAL: NCT07266363
Title: SYNERGY Study: Early Detection Through Integrated Evaluation of Cell-Free and Exosomal microRNAs for Biomarker-Guided Screening of Esophageal Squamous Cell Carcinoma
Brief Title: Integrated Cf-miRNA and Exosomal miRNA Signature for Early Detection of Esophageal Squamous Cell Carcinoma
Acronym: SYNERGY
Status: Recruiting | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 23228/SYNERGY
Record Dates: First submitted 2025-11-18; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: ESCC
Keywords: Exosomal miRNAs; Cell-free miRNAs; Esophageal squamous cell carcinoma; Liquid biopsy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — RNA from plasma or serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Discovery cohort (ESCC): Patients with ESCC
  Interventions: Diagnostic Test: Small RNA sequencing of exo- and cf-miRNAs
- Discovery cohort (NDC): Non-Disease Control
  Interventions: Diagnostic Test: Small RNA sequencing of exo- and cf-miRNAs
- Training cohort (ESCC): Patients with ESCC
  Interventions: Diagnostic Test: PCR-based validation (SYNERGY assay)
- Training cohort (NDC): Non-Disease Control
  Interventions: Diagnostic Test: PCR-based validation (SYNERGY assay)
- Testing cohort (ESCC): Patients with ESCC
  Interventions: Diagnostic Test: RT-qPCR quantification of cf- and exo-miRNAs (SYNERGY assay)
- Testing cohort (NDC): Non-Disease Control
  Interventions: Diagnostic Test: RT-qPCR quantification of cf- and exo-miRNAs (SYNERGY assay)

INTERVENTIONS:
Diagnostic Test: Small RNA sequencing of exo- and cf-miRNAs — Identification of differentially expressed cf-miRNAs
  Groups: Discovery cohort (ESCC); Discovery cohort (NDC)
Diagnostic Test: RT-qPCR quantification of cf- and exo-miRNAs (SYNERGY assay) — RT-qPCR quantification of cf- and exo-miRNAs, and construction of machine learning classifier
  Groups: Testing cohort (ESCC); Testing cohort (NDC)
Diagnostic Test: PCR-based validation (SYNERGY assay) — PCR-based validation of the SYNERGY miRNA panel
  Groups: Training cohort (ESCC); Training cohort (NDC)

SUMMARY:
Esophageal squamous cell carcinoma (ESCC) remains a highly lethal cancer worldwide, largely due to late diagnosis. Current screening methods such as upper endoscopy are invasive, operator-dependent, and limited in their ability to detect early-stage lesions.

To address this clinical need, the SYNERGY study seeks to develop a non-invasive, blood-based biomarker assay that integrates cell-free microRNAs (cf-miRNAs) and exosomal microRNAs (exo-miRNAs) to detect ESCC at an early and potentially curable stage.

This multicenter translational study includes discovery, training, and validation phases using preoperative plasma or serum samples. By combining the tumor specificity of exosomal miRNAs with the systemic sensitivity of cf-miRNAs, SYNERGY aims to construct a robust diagnostic model with high sensitivity and specificity for early ESCC detection.

DETAILED DESCRIPTION:
Esophageal cancer is the 11th most common cancer globally and the 7th leading cause of cancer-related death, with an estimated 511,000 new cases and 445,000 deaths annually. ESCC accounts for the majority of cases worldwide. Despite advances in endoscopy and therapy, outcomes for advanced ESCC remain poor, highlighting the pressing need for sensitive, minimally invasive early detection strategies.

Exosomal miRNAs (exo-miRNAs) are selectively released by tumor cells and remain stable in circulation, enabling reliable detection of tumor-specific signals. Cell-free miRNAs (cf-miRNAs) circulate broadly and can reflect overall tumor burden, metastatic spread, and microenvironmental changes.

Previous ESCC biomarker studies were limited by small validation cohorts and reliance on tissue-based public datasets that do not fully capture circulating biomarker patterns. The SYNERGY study addresses these limitations through comprehensive discovery analysis and multi-cohort blood-based validation.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 to 90 years
* Histologically confirmed esophageal squamous cell carcinoma
* No prior systemic therapy before sample collection
* For control groups: absence of malignant disease

Exclusion Criteria:

* Lack of informed consent
* Inadequate sample volume or RNA quality
* Prior cancer within 5 years (except localized cancers)
* Active systemic inflammation that may alter circulating RNA profiles

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with histologically confirmed ESCC Healthy volunteers or non-disease controls (NDC)
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2026-06-18 (Estimated); Study Completion 2026-06-18 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | At study completion, an average of one year
  Comparison of Pathological Diagnosis and the SYNERGY Assay

SECONDARY OUTCOMES:
AUC | At Study completion, an average of one year
  AUC of integrated cf- + exo-miRNA model
Specificity | Time Frame: At study completion, , an average of one year
  Description: Comparison of Pathological Diagnosis and the SYNERGY Assay

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Goel, PhD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Monrovia, California, United States

IPD SHARING:
Plan to Share IPD: No
De-identified participant data will be made available at the time of publication through a signed data access agreement, pending approval by the investigators for proposed scientific use.

REFERENCES:
- [Background] Mao Y, Fu Z, Zhang Y, Dong L, Zhang Y, Zhang Q, Li X, Wang C. A six-microRNA risk score model predicts prognosis in esophageal squamous cell carcinoma. J Cell Physiol. 2019 May;234(5):6810-6819. doi: 10.1002/jcp.27429. Epub 2018 Nov 1. PMID 30387125
- [Background] Li T, Sun G, Ye H, Song C, Shen Y, Cheng Y, Zou Y, Fang Z, Shi J, Wang K, Dai L, Wang P. ESCCPred: a machine learning model for diagnostic prediction of early esophageal squamous cell carcinoma using autoantibody profiles. Br J Cancer. 2024 Sep;131(5):883-894. doi: 10.1038/s41416-024-02781-w. Epub 2024 Jul 2. PMID 38956246
- [Background] Li K, Lin Y, Zhou Y, Xiong X, Wang L, Li J, Zhou F, Guo Y, Chen S, Chen Y, Tang H, Qiu X, Cai S, Zhang D, Bremer E, Jim Yeung SC, Zhang H. Salivary Extracellular MicroRNAs for Early Detection and Prognostication of Esophageal Cancer: A Clinical Study. Gastroenterology. 2023 Oct;165(4):932-945.e9. doi: 10.1053/j.gastro.2023.06.021. Epub 2023 Jul 1. PMID 37399999
- [Background] Miyoshi J, Zhu Z, Luo A, Toden S, Zhou X, Izumi D, Kanda M, Takayama T, Parker IM, Wang M, Gao F, Zaidi AH, Baba H, Kodera Y, Cui Y, Wang X, Liu Z, Goel A. A microRNA-based liquid biopsy signature for the early detection of esophageal squamous cell carcinoma: a retrospective, prospective and multicenter study. Mol Cancer. 2022 Feb 11;21(1):44. doi: 10.1186/s12943-022-01507-x. PMID 35148754
- [Background] Chen J, Zheng Y, Wang Z, Gao Q, Hao K, Chen X, Ke N, Lv X, Weng J, Zhong Y, Huang Z, Fu M, Zhao L, Lin F, Mi H, Tang H, Yu C, Huang Y. Development a glycosylated extracellular vesicle-derived miRNA Signature for early detection of esophageal squamous cell carcinoma. BMC Med. 2025 Jan 23;23(1):39. doi: 10.1186/s12916-025-03871-z. PMID 39849483
- [Background] Codipilly DC, Wang KK. Squamous Cell Carcinoma of the Esophagus. Gastroenterol Clin North Am. 2022 Sep;51(3):457-484. doi: 10.1016/j.gtc.2022.06.005. Epub 2022 Aug 29. PMID 36153105
- [Background] Jemal A, Bray F, Center MM, Ferlay J, Ward E, Forman D. Global cancer statistics. CA Cancer J Clin. 2011 Mar-Apr;61(2):69-90. doi: 10.3322/caac.20107. Epub 2011 Feb 4. PMID 21296855
- [Background] Codipilly DC, Qin Y, Dawsey SM, Kisiel J, Topazian M, Ahlquist D, Iyer PG. Screening for esophageal squamous cell carcinoma: recent advances. Gastrointest Endosc. 2018 Sep;88(3):413-426. doi: 10.1016/j.gie.2018.04.2352. Epub 2018 Apr 27. PMID 29709526
- [Background] Chen J, Liu X, Zhang Z, Su R, Geng Y, Guo Y, Zhang Y, Su M. Early Diagnostic Markers for Esophageal Squamous Cell Carcinoma: Copy Number Alteration Gene Identification and cfDNA Detection. Lab Invest. 2024 Oct;104(10):102127. doi: 10.1016/j.labinv.2024.102127. Epub 2024 Aug 23. PMID 39182610
- [Background] Ma L, Dou L, Liu Y, Zhang Y, Liu X, Ng HL, Chu J, Liu Y, Li Z, Ke Y, Liu S, He S, Wang G. Development and validation of predictive models combining cell-Free DNA motifs and protein biomarkers for early detection of esophageal squamous cell carcinoma and precancerous lesion. Biomark Res. 2025 Oct 14;13(1):126. doi: 10.1186/s40364-025-00840-9. PMID 41088482
- [Background] Zheng Y, Xing W, BingWei, Liu X, Liang G, Yuan D, Yang K, Wang W, Chen D, Ma J. Detection of a novel DNA methylation marker panel for esophageal cancer diagnosis using circulating tumor DNA. BMC Cancer. 2024 Dec 26;24(1):1578. doi: 10.1186/s12885-024-13301-7. PMID 39725880